CLINICAL TRIAL: NCT01619033
Title: Pharmacokinetics of 20 mg BF2.649 in Single Dose, in Subjects With Normal Renal Function Compared to Subject With Impaired Renal Function
Brief Title: Pharmacokinetics of BF2.649 in Renal Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bioprojet (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P09-13 / BF2.649; 2011-001430-42 (EudraCT Number)
Record Dates: First submitted 2011-07-20; First posted 2012-06-14 (Estimated); Last update posted 2013-04-12 (Estimated); Status verified 2013-04

CONDITIONS: Renal Impairment
Keywords: Renal impairment
MeSH Terms: conditions — Renal Insufficiency | interventions — pitolisant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- impaired renal function subjects (Experimental): impaired renal function subjects
  Interventions: Drug: BF2.649
- Healthy volunteers (Other): matched with impaired renal function subjects on ethnic group, sex, age (+/- 5 years), and BMI (+/- 20%)
  Interventions: Drug: BF2.649

INTERVENTIONS:
Drug: BF2.649 — single dose 20 mg
  Other Names: Pitolisant

SUMMARY:
This is an open, parallel group study in subjects with normal renal function compared to those with renal dysfunction.

DETAILED DESCRIPTION:
The pharmacokinetic of BF2.649 (pitolisant) is already well established from several studies in healthy human, and a recent pharmacokinetic study gave data on 12 young healthy volunteers compared to 12 elderly subject receiving 20mg/day during 14 days.

The aim of this study is to investigate effect of renal impairment on the pharmacokinetics of BF2.649 administrated on a single oral dose of 20 mg.

The once daily dose of 20 mg BF2.649 (pitolisant) chosen for this study corresponds to the usual therapeutic dose.

Twenty four subjects will be stratified according to renal function by using assessment of glomerular filtration rate (GFR) as defined by MDRD formula as follows:

* 4 subjects from 18 to 75 years of age with mild impaired renal function defined by GFR between 60 and 89 ml/min (STAGE 2 according to the international classification of chronic kidney disease)
* 4 subjects from 18 to 75 years of age with moderate impaired renal function defined by GFR between 30 and 59 ml/min (STAGE 3 according to the international classification of chronic kidney disease)
* 4 subjects from 18 to 75 years of age with severe impaired renal function defined by GFR between 15 and 29 ml/min (STAGE 4 according to the international classification of chronic kidney disease)
* 12 healthy subjects with normal renal function defined by GFR>90 ml/min with no proteinuria (<0.15g/L determined by urinalysis) matched with impaired renal function subjects on ethnic group, sex, age (+/- 5 years), and BMI (+/- 20%)

ELIGIBILITY:
Inclusion Criteria:

For subjects with impaired renal function:

* Subjects 18 to 75 years old with impaired renal function (MDRD formula between 15 and 89mL/min) medically stable since 3 months
* With body mass index (weight/height2) in the range 18 to 32 kg/m2 (inclusive)

For healthy subjects:

* Healthy subjects 18 to 75 years old with normal renal function (MDRD > 90 mL/min) and no proteinuria (<0.15g/L determined by urinalysis) matched with impaired renal function subjects on ethnic group, sex, age (+/- 5 years), and BMI (+/- 20%)

Exclusion Criteria:

For impaired renal function subjects:

* History of hepatic, cardiovascular (including conduction disturbance) or psychiatric disorder or any other condition which, in the opinion of the investigator, would jeopardize the safety of the subject or impact the validity of study results.
* Evidence of liver disease
* Presence of concomitant pathology requiring intake of any drugs or substances known to be inhibitors or inductors of CYP enzymes
* Presence of metabolic or ionic disorders not controlled by adapted treatment
* Presence of significant anemia,nephrotic syndrome
* Renal transplantation

For healthy subjects:

* history of renal, cardiovascular, gastrointestinal, hepatic, neurological, endocrine or psychiatric disorders or any surgery which puts them at risk in the opinion of the investigator.
* Any treatment within 14 days before inclusion, or within 5 times the elimination half-life of that drug, whichever the longest, including treatment which could lead to inhibition or induction of CYP enzymes - mainly CYP3A4 and CYP2D6 and with the exception of hormonal contraception and menopausal hormone replacement therapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2011-07; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Mesure of classic pharmacokinetic parameters determined on BF2.649 serum and urine concentration | between H0(0hr - Pre-dose) and H96 (96hr) after single oral dose
  Cmax, Tmax, AUClast, AUC∞, λz, t½term, CL/F, Vz/F

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | during the 4 days following the drug administration
  clinical safety of BF2.649.
change in lab tests (biological and clinical safety) | during 4 days after drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Claire POUTEIL-NOBLE, MD, Principal Investigator — Nephrologie, Centre Hospitalier Lyon Sud
Locations (1):
- EUROFINS OPTIMED Lyon, Lyon, France